CLINICAL TRIAL: NCT02495246
Title: A Phase I, Safety and Immunogenicity Trial of the Heterologous Prime-boost Regimen Combining the Monovalent Zaire Ebola Viral Vector Candidates ChAd3-EBO-Z and Ad26.ZEBOV in Healthy UK Adults
Brief Title: A Study to Assess Ebola Vaccines ChAd3-EBO-Z and Ad26.ZEBOV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EBL05
Record Dates: First submitted 2015-06-18; First posted 2015-07-13 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

ARMS (4):
- Group 1 (Active Comparator): ChAd3-EBO-Z (1x10^11 vp) and Ad26.ZEBOV (5x10^10 vp) 28 days later.
  Interventions: Biological: ChAd3-EBO-Z; Biological: Ad26.ZEBOV
- Group 2 (Active Comparator): Ad26.ZEBOV (5x10^10 vp) and ChAd3-EBO-Z (1x10^11 vp) 28 days later.
  Interventions: Biological: ChAd3-EBO-Z; Biological: Ad26.ZEBOV
- Group 3 (Active Comparator): ChAd3-EBO-Z (1x10^11 vp) and Ad26.ZEBOV (5x10^10 vp) 56 days later.
  Interventions: Biological: ChAd3-EBO-Z; Biological: Ad26.ZEBOV
- Group 4 (Active Comparator): Ad26.ZEBOV (5x10^10 vp) and ChAd3-EBO-Z (1x10^11 vp) 56 days later.
  Interventions: Biological: ChAd3-EBO-Z; Biological: Ad26.ZEBOV

INTERVENTIONS:
Biological: ChAd3-EBO-Z
Biological: Ad26.ZEBOV

SUMMARY:
This is a clinical trial in which healthy volunteers will be administered two experimental Ebola vaccines: ChAd3-EBO-Z and Ad26.ZEBOV. Four groups of volunteers will be vaccinated with both vaccines one after the other in a prime/boost regimen.

All ChAd3-EBO-Z doses are 1x10^11 vp and all Ad26.ZEBOV doses are 5x10^10 vp.

Group 1 will receive a ChAd3-EBO-Z priming vaccine and an Ad26.ZEBOV boosting vaccine 28 days later.

Group 2 will receive an Ad26.ZEBOV priming vaccine and a ChAd3-EBO-Z boosting vaccine 28 days later.

Group 3 will receive a ChAd3-EBO-Z priming vaccine and an Ad26.ZEBOV boosting vaccine 56 days later.

Group 4 will receive an Ad26.ZEBOV priming vaccine and a ChAd3-EBO-Z boosting vaccine 56 days later.

The study will assess the safety of the vaccinations, and the immune responses to vaccination. Immune responses are measured by tests on blood samples.

The ChAd3-EBO-Z and Ad26.ZEBOV vaccines are called viral vectored vaccines. They are made from viruses which are modified so that they cannot multiply. The viruses have extra DNA in them so that after injection, the body makes Ebola proteins (but Ebola does not develop), so that the immune system builds a response to Ebola without having been infected by it.

Healthy volunteers will be recruited in Oxford and London, England. The study will be co-funded by GSK Biologicals and Crucell Holland BV.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss the volunteer's medical history with their GP
* For females only, willingness to practice continuous effective contraception (see section 6.3.3) during the study and a negative pregnancy test on the day(s) of screening and vaccination
* Agreement to refrain from blood donation during the course of the study
* Provide written informed consent

Exclusion Criteria:

* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational Ebola or Marburg vaccine, a chimpanzee adenovirus, or any other investigational vaccine likely to impact on interpretation of the trial data
* Receipt of any live, attenuated vaccine within 28 days prior to enrolment
* Receipt of any subunit or killed vaccine within 14 days prior to enrolment
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, (e.g. egg products) including urticaria, respiratory difficulty or abdominal pain
* Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
* Any history of anaphylaxis in reaction to vaccination
* Pregnancy, lactation or willingness/intention to become pregnant during the study
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition
* Poorly controlled asthma or thyroid disease
* Seizure in the past 3 years or treatment for seizure disorder in the past 3 years
* Bleeding disorder (eg. Factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
* Any other serious chronic illness requiring hospital specialist supervision
* Current anti-tuberculosis prophylaxis or therapy
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the 5 years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Travel to a Ebola or Marburg endemic region during the study period or within the previous six months
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis (see Appendix A and Appendix B)
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of administration of ChAd3-EBO-Z and Ad26.ZEBOV 28 days later. This will be done by recording the number of participants who experience adverse events and the severity of any adverse events. | 17 weeks
Safety and tolerability of administration of Ad26.ZEBOV and ChAd3-EBO-Z 28 days later. This will be done by recording the number of participants who experience adverse events and the severity of any adverse events. | 17 weeks
Safety and tolerability of administration of ChAd3-EBO-Z and Ad26.ZEBOV 56 days later. This will be done by recording the number of participants who experience adverse events and the severity of any adverse events. | 21 weeks
Safety and tolerability of administration of Ad26.ZEBOV and ChAd3-EBO-Z 56 days later. This will be done by recording the number of participants who experience adverse events and the severity of any adverse events. | 21 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Oxford, Oxfordshire, United Kingdom